CLINICAL TRIAL: NCT03339986
Title: Manipulation of Snack Intake in Young Children Using Snack Replacement and Snack Reduction
Brief Title: Downsizing: Snacking in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sophie Reale (Other)
Collaborators: University of Leeds (Other); University of St Andrews (Other)
Responsible Party: Sponsor-Investigator, Sophie Reale, PhD student, University of Sheffield
Organization: University of Sheffield (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 007850
Record Dates: First submitted 2017-08-23; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Food Habits; Food, Snack; Acceptance Processes
Keywords: Portion Size; Feasibility; Acceptability; Snacking; Preschool children
MeSH Terms: conditions — Feeding Behavior; Behavior | interventions — Replantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduction (Experimental): Participants will be instructed to reduce all high energy dense snacks that they serve to thier children by 50%
  Interventions: Behavioral: Reduction or Replacement
- Replacement (Experimental): Participants will be instructed to replace all high energy dense snacks with fresh fruit and vegetables
  Interventions: Behavioral: Reduction or Replacement

INTERVENTIONS:
Behavioral: Reduction or Replacement

SUMMARY:
The aim of the study is to investigate and compare two strategies of portion control in toddlers aged 24 to 59 months (snack replacement and snack reduction). The investigators aim to compare the effect of these strategies on habitual dietary intake (total energy intake (kcal), sugar intake (g), intake of fruits and vegetables, and intake at a test meal provided in the home (total energy intake (kcal) and intake of each component of the meal, e.g. intake of vegetables). Outcome measures will be compared to baseline within strategies and also between strategies to explore which portion control strategy might be most effective.

DETAILED DESCRIPTION:
Following provision of informed consent the primary caregiver will be provided with a recruitment questionnaire. The questionnaire can be completed on paper or online (identical questionnaires). It will include the Food Frequency Questionnaire (FFQ; Hammond et al., 1993) to determine whether the child likes and regularly eats HED snacks. A FFQ will also be administered to the main caregiver in order to establish familial patterns of food intake.

Demographic information will be collected for both caregivers and child in paper or online format. Measures of child eating behaviour, parental feeding practices, food neophobia and temperament will be taken. Anthropometric information of the child will also be collected by the researcher to calculate weight-for-height z scores.

A between-subject 3-week intervention will be implemented with participants acting as their own controls during the baseline (week 1) and acclimation (week 2) periods before being randomised in to the intervention period (week 3) (figure 1). Caregivers will be instructed to complete a 4-day weighed food diary each week (3 weekdays and at least one weekend day). This will involve the caregiver recording all food and drinks consumed by their child to the nearest gram using the scales provided.

During week 1 (baseline) parents will be instructed to make no alterations to the foods and drinks that they provide to their child. Data from this phase of the experiment will be used to examine the habitual diet. Data obtained in this phase will enable us to determine whether or not the provision of the snacks has changed the child's dietary habits.

During week 2 (acclimation phase) participants will be provided with a range of snacks that are intended to replace all usual snacks. This will consist of several different snack options (figure 2) to provide up to three snacks per day and to allow for any siblings who may want an identical snack option. All participants will be provided with the same selection of HED snacks, which will be familiar to all children. Snack types and amounts will be based on data collected from the cohort prior to the beginning of the experiment when participants express an interest in taking part. Parents/ caregivers will be required to replace all usual snacks with the ones provided over the following 7 days and will be instructed to provide the snacks at their child's usual snack time following a snacking schedule, and to record it in the food diary; this will allow the snacking schedule to be matched in week three. If parents usually provide fruit or vegetables (in their natural form) for a snack occasion they will be instructed to continue to do so. HED snacks are being provided in this pilot study to ensure consistency across all children.

In week 3 parents will be randomly allocated (block randomisation) to one of two portion size reduction interventions via simple randomisation procedure (snack reduction or snack replacement). Caregivers will be instructed to either reduce all snacks by 50% or replace all snacks with familiar and relatively liked fruits, vegetables and a starch component (breadstick, cracker or rice cake). In the snack reduction condition parents and caregivers will be provided with the same snacks as in week 2 and a snacking schedule showing the amounts and types of snacks that should be offered to the child (as per week 2). Once the downsized snack (50% portion) has been consumed, if the child indicates that they are still hungry, caregivers will be advised to offer any other low energy dense foods such as fruits and vegetables. In the replacement condition, caregivers will be instructed to remove all HED snacks that were provided in week 2 or otherwise and sugar sweetened beverages from the child's diet for one week and offer only the fruits and vegetables, starch-based food (bread stick, rice cake or cracker) and sugar free drinks provided. All participants in the snack replacement group will be provided with a snack pack consisting of fruits and vegetables familiar and relatively liked to all children (for example apples, grapes, pears, banana, red pepper, cucumber, cherry tomatoes and carrots (all served raw)). The fruit and vegetable types will be based on the data collected on children familiarity of fruits and vegetables from the cohort prior to week 1.Caregivers will be instructed to offer 40g of both a specified fruit and vegetable (more if the child requests) and a pre-defined starch component. This is based on a typical portion size for a pre-school child. A snacking schedule will also be provided for the fruits and vegetables.

ELIGIBILITY:
Inclusion Criteria:

* Parents/ caregivers of children aged 24-59 months old
* Must consume a HED snack at least once per day.
* Written informed consent provided from caregivers/ parents.

Exclusion Criteria:

* Children who attend nursery for more than three full consecutive days will be excluded due to the requirement of a four-day consecutive food diary to be completed in the home environment.
* Children with food allergies, long-term health conditions known to affect food intake, who are taking medication known to affect appetite, and those who report dislike of the snacks provided will be excluded from taking part.
* Children whose parents report a dislike of the study foods will also be excluded from taking part in the study.
* Children whose parents report no commercially available snack intake will be excluded from taking part in the study since participants will be required to reduce their children's snack intake by 50% or replace it with a LED alternative. At least one high energy dense, commercially available snack (e.g. chocolate, crisps) must normally be consumed per day by the child
* Parent child pairs must be able to commit to three consecutive weeks in order to take part in the study.
* Participant who are excluded from taking part in the current study will be invited to take part in our future studies where no study food will be provided.

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2017-08-12 (Actual)

PRIMARY OUTCOMES:
Retention | 9 months
  The number of people that adhered to the protocol

SECONDARY OUTCOMES:
Participation | 9 months
  The number of days each participant complied to the snacking schedule
Acceptability | 9 months
  A score derived from a 15 item questionnaire
Preliminary effects of the intervention | 9 months
  Energy intake (kcal)
Preliminary effects of the intervention | 9 months
  Sugar intake (grams)
Preliminary effects of the intervention | 9 months
  Salt intake (grams)
Preliminary effects of the intervention | 9 months
  Fat intake (grams)
Preliminary effects of the intervention | 9 months
  Fruit intake (grams)
Preliminary effects of the intervention | 9 months
  Vegetable intake (grams)
Sustainability of effect | 9 months
  Frequency of consumption (FFQ)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha J Caton, PhD, Principal Investigator — University of Sheffield

IPD SHARING:
Plan to Share IPD: No